CLINICAL TRIAL: NCT01046981
Title: Tumescent Antibiotic Delivery: Pharmacokinetic Evidence for Improved Surgical Site Infection Prevention
Brief Title: Tumescent Antibiotic Delivery Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Klein, Jeffrey A., M.D. (Individual)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2 TAD
Record Dates: First submitted 2010-01-11; First posted 2010-01-12 (Estimated); Last update posted 2011-09-28 (Estimated); Status verified 2011-09

CONDITIONS: Prevention of Surgical Site Infections
Keywords: Surgical site infections; Prevention; Prophylaxis; Tumescent; Intravenous; Antibiotic; Absorption; Pharmacokinetics; Bioavailability
MeSH Terms: conditions — Surgical Wound Infection | interventions — Metronidazole; Cefazolin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tumescent Antibiotic Delivery (Experimental): TAD followed by sequential serum and interstitial tissue fluid sampling for antibiotic concentration of subsequent 24 hours
  Interventions: Procedure: Tumescent Antibiotic Delivery of cefazolin with or without metronidazole
- Intravenous Antibiotic Delivery (Experimental): Intravenous antibiotic delivery of cefazolin with or without metronidazole followed by sequential serum and interstitial tissue fluid sampling for antibiotic concentration of subsequent 24 hours.
  Interventions: Procedure: Intravenous Antibiotic Delivery

INTERVENTIONS:
Procedure: Tumescent Antibiotic Delivery of cefazolin with or without metronidazole — TAD of cefazolin with or without metronidazole followed by sequential serum and interstitial fluid samples over 14 to 24 hours for antibiotic concentrations
  Other Names: Cefazolin; Metronidazole
  Arms: Tumescent Antibiotic Delivery
Procedure: Intravenous Antibiotic Delivery — Intravenous antibiotic delivery of cefazolin with or without metronidazole followed by sequential serum sampling for antibiotic concentration of subsequent 12 to 24 hours.
  Arms: Intravenous Antibiotic Delivery

SUMMARY:
Tumescent Antibiotic Delivery (TAD) is a technique for improving the prevention of surgical site infections (SSI). TAD involves the subcutaneous infiltration of tumescent local anesthesia (TLA) containing water soluble antibiotic(s) such as cefazolin and metronidazole. TLA consists of the subcutaneous infiltration of very dilute lidocaine (≤ 1 gram/liter) and epinephrine (≤ 1 milligram/liter) with sodium bicarbonate (10 milliequivalents/liter) in a physiologic solution of sodium chloride which produces intense local anesthesia associated with profound wide-spread vasoconstriction lasting for more than 12 hours. Compared to intravenous antibiotic delivery (IVAD), TAD is expected to produce higher local tissue concentrations of the antibiotic(s) for longer periods of time and lower systemic/serum antibiotic concentrations. This clinical trial will compare TAD to IVAD with respect to pharmacokinetic evidence for possible improved SSI prevention.

DETAILED DESCRIPTION:
The protocol entitled Absorption Kinetics of Subcutaneous Tumescent Cefazolin and Metronidazole is a Phase I dose ranging clinical study designed to document the concentration-time profile of cefazolin and lidocaine after subcutaneous infiltration of cefazolin in tumescent local anesthesia (TLA). The antibiotic cefazolin is routinely given intravenously (IV) for the prophylaxis of surgical site infections (SSI).

Tumescent local anesthesia (TLA) consists of the subcutaneous infiltration of very dilute lidocaine (≤ 1 gram/liter) and epinephrine (≤ 1 milligram/liter) with sodium bicarbonate (10 milliequivalents/liter) in a physiologic solution of sodium chloride. Clinically TLA produces intense local anesthesia associated with profound wide-spread vasoconstriction lasting for more than 12 hours. Tumescent delivery of a cefazolin refers to the subcutaneous infiltration of cefazolin dissolved in a dilute solution of tumescent local anesthesia.

For a number of surgical procedures the current standard of care for prophylaxis of surgical site infection (SSI) is IV antibiotics (e.g. cefazolin) administered within 30 to 60 minutes before a surgical incision. We hypothesize that tumescent delivery of cefazolin may be more effective in preventing SSI and possibly safer with fewer side effects compared to IV delivery of cefazolin.

This protocol is a preliminary step in exploring the possibility that tumescent delivery of cefazolin is better than standard IV delivery for the prevention of SSI. The present protocol is a phase I study that will document and compare serum and tissue cefazolin levels after IV and subcutaneous tumescent delivery. A finding that tumescent delivery provides prolonged tissue levels of cefazolin will justify a phase II study of tumescent cefazolin at the site of an anticipated surgical incision for SSI prevention.

• Summary of Experimental Design of Clinical Trial Protocol The tumescent cefazolin study protocol is organized as follows. The tumescent cefazolin clinical study protocol will involve four adult volunteer subjects/participants. Each subject will participate in up to four (4) separate 12 to 24-hour investigative procedures at least one to two weeks apart. Concentrations of drugs in the solution of tumescent local anesthesia will be: lidocaine ≤ 1000 mg/L, epinephrine ≤ 1.0 mg/L, sodium bicarbonate 10 meq/L, cefazolin ≤ 1 gm/L with or without metronidazole 500mg/L . Maximum total cefazolin dose will be 1 gm. The maximum total metronidazole dose will be 500 mg. The maximum tumescent lidocaine dosage will be 20 mg/kg. TLA will be delivered into subcutaneous fat by peristaltic infiltration pump using blunt-tipped infiltration cannulas.

Procedures 1 & 2: Subcutaneous infiltration of tumescent cefazolin: Two of the four investigative procedures will begin with infiltration of a solution of tumescent local anesthesia containing cefazolin. Following infiltration of subcutaneous tumescent local anesthesia containing cefazolin approximately 9 sequential blood and tissue samples are taken over 12 to 24 hours. In these two studies a minimal volume of liposuction (10 ml to 12 ml using a hand held syringe) will be done in order to obtain samples of subcutaneous fat and tumescent subcutaneous interstitial tissue-fluid for measurement of cefazolin and metronidazole concentration.

Procedure 3: IV infusion of cefazolin or metronidazole: In the control study the patient is given 1 gm of IV cefazolin with or without 500 mg of metronidazole and subsequent sequential serum samples for antibiotic concentration will be obtained over 12 hours.

Serum Samples: Sequential sampling of serum and fat will be obtained at 0, 1, 3, 6, 9, 12, 18, and 24 hour (T0, T1, T3, T6, T9, T12, T15, T18 and T24), where T0 = time of completion of tumescent infiltration or IV infusion. Serum samples will be obtained from a peripheral vein via an indwelling catheter and analyzed for cefazolin concentration by HPLC.

Tissue Fluid Samples: Samples of subcutaneous tissue fluid will be obtained by liposuction of approximately 10 ml of subcutaneous fat and tumescent anesthetic solution using a hand-held syringe, the aspirate being centrifuged to obtain an aqueous infranate from which cefazolin, metronidazole and lidocaine concentration will be measured by HPLC. Clinical experience has shown that tumescent local anesthesia persists for at least 12 hours. If the patient experiences any significant discomfort during the aspiration of subcutaneous fat using a hand-held syringe, then no further subcutaneous tissue samples will be taken for the duration of that clinical procedure.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult
* No allergies to cefazolin, metronidazole or lidocaine

Exclusion Criteria:

* HIV
* Hepatitis C
* Diabetes

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2009-03; Primary Completion 2011-04 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve (AUC) of antibiotic concentration as a function of time | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Capistrano Surgery Center, San Juan Capistrano, California, United States

REFERENCES:
- See also: Information about tumescent drug delivery — http://www.tumescent.org